CLINICAL TRIAL: NCT05179252
Title: POD and Postoperative Outcomes in Senile Patients After SFI for Hip Fracture Surgery: A Randomized Trial
Brief Title: Shenfu Injection for Postoperative Delirium (SFI for POD)
Acronym: POD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong University of Traditional Chinese Medicine (Other)
Collaborators: Shandong Institute of Science and Technology Information (Other)
Responsible Party: Principal Investigator, weiliang zhang, Principal Investigator, Shandong University of Traditional Chinese Medicine
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SZYA20210603-A1
Record Dates: First submitted 2021-11-16; First posted 2022-01-05 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-12

CONDITIONS: Postoperative Delirium
MeSH Terms: conditions — Emergence Delirium | interventions — Shen-Fu; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SFI intervention group (Experimental): shenfu injection used during surgery, day one and two after surgery, 50ml,iv drop.
  Interventions: Drug: Shen-Fu injection
- Control group (Sham Comparator): same volume of normal saline used during surgery, day one and two after surgery, 50ml,iv drop.
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Shen-Fu injection — Chinese patent medicine made by modern technology
  Other Names: sanjiu yaan
  Arms: SFI intervention group
Drug: normal saline — 0.9% normal saline, used for sham control
  Other Names: physiological saline solution
  Arms: Control group

SUMMARY:
Surgery or trauma may cause serious problem to patients, especially for senile ones, like postoperative delirium or more postoperative complications. Here, we conduct a investigation of SFI for preventing the happening of POD or postoperative complications.

DETAILED DESCRIPTION:
SFI(Shenfu Injection), a historical medical herbal medicine of traditional Chinese, which may produced much benefit to clinical patients with furtigue after major surgery, because it was a comment sense to think of energy loss if they experience surgical damage. Here, we administrated intravenously SFI into senile patients, who receiving hip fracture surgery, to avoid bad results or serious postoperative outcomes, in case of enhancing recovery after surgery.

ELIGIBILITY:
Inclusion Criteria:

* hip fracture surgery under epidural anesthesia

Exclusion Criteria:

* Severe dementia, hearing/vision impairment, coma, etc., unable to communicate;
* patients with end-stage diseases such as tumor;
* 3 months after myocardial infarction, cerebral infarction;
* severe heart, liver and renal dysfunction.

Ages: 75 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
incidence of postoperative delirium within 7 days | day 1-7 after surgery, more scores means higher incidence of POD
  postoperative delirium(POD), assessed with Confusion Assessment Method scale and Richmond Agitation-Sedation Scale together.

SECONDARY OUTCOMES:
non-delirium complications | day 1-7 after surgery
  postoperative complications except for delirium
length of stay | approximately day 1 in hospital to day 7
  length of hospital stay
pain assessment within 3 days | day 1-3 after surgery, higher scores mean more pain.
  postoperative pain estimated with Numerical Rating Scale
all-caused mortality within 30 days | 30 days after surgery
  short-term follow up
survival in 1 year | 1 year discharge from hospital
  long-term follow up
adverse events to shenfu injection | approximately day1-7 after surgery
  adverse events caused form shenfu injection

CONTACTS AND LOCATIONS:
Overall Officials: zhang xin, Study Director — Shandong University of Traditional Chinese Medicine

IPD SHARING:
Plan to Share IPD: No